CLINICAL TRIAL: NCT07350291
Title: Evaluation of the Diagnostic Capabilities of Saliva Samples From Pediatric Patients, Promoting Active Involvement of the Individuals Concerned and Their Families: Protocol for a Randomized Intra-individual Study.
Brief Title: Evaluation of the Diagnostic Capabilities of Saliva Samples From Pediatric Patients, Promoting Active Involvement of the Individuals Concerned and Their Families.
Acronym: Presap
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Presap; PHRIP (Other Grant/Funding Number: DGOS ministère de la santé)
Record Dates: First submitted 2025-12-31; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Pediatrics; Virus Diseases in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm with nasopharyngeal suction (Active Comparator): This stand sample is the current gold standard for collecting winter virii in paediatrics. It consists of aspirating serosities via a nasopharyngeal device.
  Interventions: Diagnostic Test: The aim is to compare the effectiveness of virological and bacterial detection between two sampling methods
- Experimental arm with nasopharyngeal swab (Experimental): This experimental sample will consist of inserting a weighted dummy into the oral cavity, in order to obtain a sample of the child's saliva and compare it with the standard sample.
  Interventions: Diagnostic Test: The aim is to compare the effectiveness of virological and bacterial detection between two sampling methods

INTERVENTIONS:
Diagnostic Test: The aim is to compare the effectiveness of virological and bacterial detection between two sampling methods — The nasopharyngeal swab and the buccal swab will be taken separately as a cross over with randomisation carried out to allow a different order for each patient. The collection time, the quantity of virus, the quality of the sample and the human intervention will be quantified.The pain and comfort of both carers and children will be assessed.
  Other Names: standard; experimental

SUMMARY:
The management of respiratory infections accounts for a large proportion of winter activity in paediatric wards. The main pathologies are bronchiolitis, affecting infants under the age of 2. Today, the reference method for diagnosing respiratory pathogen infections is nasopharyngeal aspirate (NPA), performed by paramedical staff. However, this technique is invasive and traumatic for paediatric patients. During the SARS-CoV-2 pandemic, salivary sampling was used on a large scale in the paediatric population, and showed good concordance with reference samples, as well as better tolerance/acceptability. The aim of the PreSaP (Paediatric Saliva Sampling) study is to assess the diagnostic capabilities of saliva samples¹ . This will be a monocentric, intra-individual, randomised study involving 502 children using the results of nasopharyngeal aspirates as the gold standard. We will also evaluate the time required to take nasopharyngeal aspirates and saliva samples in order to examine any difficulties associated with the two sampling methods. Although the results of our study report few diagnostic errors, they would justify the use of saliva sampling in routine care to reduce stressful and painful factors, and thus contribute to the well-being of infants and children. Saliva sampling could improve acceptance by the child and those around him, avoiding a less negative experience while guaranteeing a reliable diagnosis of respiratory pathogens. This new technique should also encourage the active involvement of all those involved in care.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged between 28 days and under 24 months.

  * Admission to paediatric A&E or general paediatrics.
  * Respiratory conditions requiring treatment for microbiological diagnosis by upper airway sampling.
  * Collection of consent signed by legal representatives or guardians with parental authority. Except in cases where there is a single parent with parental authority.
  * Persons affiliated with or beneficiaries of a social security scheme.

Exclusion Criteria:• Refusal to participate by one of the legal representatives or the patient.

* Patients with a contraindication to ASNA (those with haemophilia, on anticoagulants or with thrombocytopenia).
* Patients with a known increased risk of epistaxis (nosebleeds), hypertrophic rhinitis or other conditions causing excessive mucosal fragility.
* Participation in another study that would impact the primary objective of this research.
* Patients who may be allergic to the material used in the sponge pacifier.
* Patients in a life-threatening emergency situation.

Ages: 28 Days to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 502 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of patient with a detection of respiratory pathogens | Day 1
  This intra-individual trial (cross-over trial where two samples are taken from each child) aims to assess the ability of a test to detect respiratory pathogens from a saliva sample, using nasopharyngeal aspiration (NPA) as the gold standard.

IPD SHARING:
Plan to Share IPD: No